CLINICAL TRIAL: NCT04369911
Title: Acupuncture Treatment for Chronic Post-traumatic Headache in Individuals With Mild Traumatic Brain Injury
Brief Title: Acupuncture in Traumatic Brain Injury
Acronym: AccuTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Minnesota Office of Higher Education (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A19-094
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2023-12

CONDITIONS: Chronic Post-traumatic Headache; Mild Traumatic Brain Injury
Keywords: acupuncture
MeSH Terms: conditions — Brain Concussion | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose (Experimental): Acupuncture treatment once per week for 5 weeks. Five total acupuncture treatments completed.
  Interventions: Procedure: Acupuncture
- High Dose (Experimental): Acupuncture treatment twice per week for 5 weeks. Ten total acupuncture treatments completed.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatments will be separated by a minimum of two days and a maximum of 14 days. Treatment sessions will be identical for both groups. Standard, sterile stainless-steel, disposable needles will be inserted at acupuncture points with a total of 18 needles for each treatment session. The depth of the needle will be approximately 10-20 millimeters. Needles will be left in place for 30 minutes.

SUMMARY:
The purpose of the study is to determine the effect of a low vs. high dose of acupuncture treatment in individuals with chronic post-traumatic headache (CPTH). A total of 36 people with mild traumatic brain injury (mTBI) suffering from CPTH will be enrolled in this study to receive acupuncture treatment for 5 weeks. Participants will be randomized into two groups: 1) Low Acupuncture group (5 treatments) and 2) High Acupuncture group (10 treatments). It is hypothesized that both treatment groups will have decreased headaches, but that 10 treatments will greater alleviate headaches when compared to 5 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide and provision of signed and dated informed consent form
* Age 18-65
* Diagnosis of mild traumatic brain injury (mTBI) (as defined by the International classification of headache disorders 3rd edition (ICHD-3); a. Either no loss of consciousness, or loss of consciousness of <30 minutes duration, b. Glascow Coma Scale (GCS) ≥ 13, and c. Symptoms and/or signs diagnostic of concussion)
* Diagnosis of mTBI ≥3 months and ≤12 months at the time of study enrollment
* Suffering from chronic post-traumatic headache (CPTH) of any etiology (e.g. tension or migraine), with chronic defined as developed within 7 days after injury and lasting ≥3 months from the time of injury
* Stable medication regimen for ≥1 months and agree to adhere to his or her current medication treatment regimen through study participation

Exclusion Criteria:

* Non-English speaking
* History of acupuncture since diagnosis of mTBI
* History of pre-existing primary headache, defined as more than 12 days of tension-type headache annually and/or more than one migraine attacks per month in the last year
* History of any other serious neurological, psychiatric, chronic pain disorders, or seizures
* History of bleeding diathesis, other bleeding disorders, or syncope with needle puncture
* History of cardiac arrhythmia or current pacemaker, neurostimulator, or other implanted stimulation device
* Recent or active substance use disorder
* Women who are currently pregnant, lactating, or planning to become pregnant during the study
* Any other medical conditions that could affect their ability to participate in acupuncture treatments for the study duration (as determined by study investigators)
* Active participation or past participation ≤3 months in any other interventional study.
* Unwilling to participate in all study related activities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda A Herrmann, PhD, Principal Investigator — HealthPartners Neuroscience Research
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was withdrawn for eligibility reasons prior to randomization to study group. This participant was not included in analysis.
Period: Overall Study
Arm/Group | Low Dose | High Dose
Started | 18 | 20
Completed | 14 | 15
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 3 | 8
  Between 18 and 65 years | 12 | 17 | 29
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (14) | 47 (12) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 20 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 12 | 17 | 29
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Time to diagnosis of TBI [Mean (Inter-Quartile Range); unit: months] | 7.5 [5.2 to 11.3] | 8.9 [4.8 to 12.9] | 7.7 [5.0 to 11.5]

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Headache Days
Description: The number of self-reported headache days over a 4 week period. Range: 0-28 days. More headache total days indicates a worse outcome.
Time Frame: baseline to 3 months
Measure: Mean (Standard Deviation); unit: headache days
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 18 | 20
headache days | -8 (10) | -6 (8)

2. Secondary Outcome: Adverse Events
Description: The total number of adverse events (AE) or serious adverse events (SAE) over the course of the study. A higher number of AE/SAEs indicates a less safe treatment.
Time Frame: 16 weeks
Measure: Number; unit: total number of AEs
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 18 | 20
total number of AEs | 13 | 25

3. Secondary Outcome: Compliance With Overall Protocol
Description: Completion of treatment sessions. Percent of target treatments. Range: 0-100. A higher percentage indicates more compliance.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of treatments completed
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 18 | 20
percentage of treatments completed | 95 (19) | 91 (27)

4. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI contains questions about participant's sleeping habits. Range: 0-21. Sum of 7 subscores. Higher score indicates worse sleep quality
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
score on a scale | 9.9 (5.0) | 9.1 (3.4)

5. Other Pre Specified Outcome: Traumatic Brain Injury-Quality of Life Headache Pain (TBI-QOL-Headache)
Description: The TBI-QOL-Headache contains questions about participant's headache pain. Raw Score Range: 10-50. Raw scores converted to T-score (mean = 50, standard deviation = 10). Higher T-score indicates more headache pain.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
T-score | 59 (5) | 58 (6)

6. Other Pre Specified Outcome: Change in Headache Pain Intensity
Description: The headache pain intensity is self reported for each headache day. Pain intensity will be averaged for the 4 week period measured. Pain intensity scale range is 0 (no pain) to 10 (worst pain imaginable). Higher pain intensity score indicates more intense headaches.
Time Frame: baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 18 | 20
score on a scale | -.57 (.74) | -.20 (1.09)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 14/18 | 17/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=18) | High Dose (N=20)
Lightheaded/Syncope (Ear and labyrinth disorders) | 2 (2) | 5 (6)
Skin Reaction at site (Skin and subcutaneous tissue disorders) | 4 (5) | 9 (18)
Skin or other issues away from site (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Pain (Musculoskeletal and connective tissue disorders) | 13 (23) | 11 (25)
Breathing issues (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Heart issues (Cardiac disorders) | 1 (1) | 0 (0)
Flu (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (Injury, poisoning and procedural complications) | 0 (0) | 3 (5)
Acute Illness (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT04369911/Prot_SAP_000.pdf